CLINICAL TRIAL: NCT00163748
Title: A Pilot Study of Outpatient Vinorelbine and Gemcitabine With Filgrastim Support for Patients With Relapsed or Refractory Lymphoma.
Brief Title: Efficacy and Treatment Related Toxicity Study of a New Regimen for Lymphoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Bayside Health (Other Government)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AH152/00
Record Dates: First submitted 2005-09-12; First posted 2005-09-14 (Estimated); Last update posted 2016-01-08 (Estimated); Status verified 2016-01

CONDITIONS: Non-Hodgkin's Lymphoma; Hodgkin's Disease
Keywords: Lymphoma
MeSH Terms: conditions — Lymphoma, Non-Hodgkin; Hodgkin Disease; Lymphoma | interventions — Gemcitabine; Vinorelbine

INTERVENTIONS:
Drug: gemcitabine, vinorelbine

SUMMARY:
This is an open label pilot study of 40 evaluable patients receiving vinorelbine-gemcitabine combination chemotherapy with filgrastim support in an outpatient setting. Participating patients at the time of registration will have measurable relapsed or primary refractory lymphoma.

DETAILED DESCRIPTION:
Patients suffering from lymphoma (a type of cancer of the white blood cells called lymphocytes) have less chance of cure if they are refractory to initial chemotherapy or relapse after receiving initial chemotherapy when compared to patients who are responsive to and do not relapse following initial chemotherapy. The standard of care, therefore, for these patients is to undergo some form of bone marrow transplant procedure. However, before this can be considered most patients require chemotherapy to control the lymphoma and to determine whether the lymphoma is still sensitive to alternative types of chemotherapy (salvage chemotherapy). Currently used types of salvage chemotherapy require significant periods of inpatient hospitalisation and are associated with significant haematological toxicities (low blood counts with the associated risks of infection and bleeding and the need for blood and platelet transfusions). Two new chemotherapy drugs, vinorelbine and gemcitabine, have both shown encouraging efficacy against lymphoma when used alone for patients with heavily pretreated lymphoma. Furthermore, they can be given in an outpatient setting and are usually not associated with significant haematological toxicity. All the patients participating in this study have been diagnosed with relapsed or refractory lymphoma and have been offered treatment with vinorelbine and gemcitabine as an alternative to inpatient salvage chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

* age 18 to 70 years
* relapsed or primary refractory non-Hodgkin's lymphoma (NHL) or Hodgkin's Disease (HD)
* measurable disease (clinically or radiologically)
* ECOG 0 - 2
* written informed consent

Exclusion criteria:

* bilirubin > 50μmol/litre unless secondary to lymphoma
* creatinine > 2 x upper limit of normal unless secondary to lymphoma,
* absolute neutrophil count <0.5 x 109/litre and / or platelets < 50 x 109/litre unless secondary to lymphoma
* isolated bone marrow disease
* known sensitivity to E coli derived preparations

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40
Dates: Start 2001-02; Primary Completion 2003-11 (Actual); Study Completion 2003-11 (Actual)

PRIMARY OUTCOMES:
To evaluate the efficacy and regimen related toxicity of the study treatment (vinorelbine and gemcitabine with filgrastim support).

SECONDARY OUTCOMES:
To evaluate the requirement for inpatient admission and / or parenteral antibiotic therapy following study treatment in an outpatient setting.

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Spencer, Assoc. Prof, Study Chair
Locations (2):
- Australia (2):
  - Royal North Shore Hospital, Sydney, New South Wales
  - The Alfred Hospital, Melbourne, Victoria